CLINICAL TRIAL: NCT00695253
Title: Physician-Sponsored IDE for Talent Endoluminal Spring Graft System in Patients With AAA
Brief Title: Physician-Sponsored IDE for Talent Endoluminal Spring Graft System in Patients With Abdominal Aortic Aneurysms (AAA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rodney A. White, M.D. (Other)
Responsible Party: Sponsor-Investigator, Rodney A. White, M.D., Chief, Vascular Surgery, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Organization: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10807-01
Record Dates: First submitted 2007-12-28; First posted 2008-06-11 (Estimated); Results first posted 2021-09-29 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Abdominal Aortic Aneurysms
Keywords: AAA
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Talent Endoluminal Spring Graft System (Other): Single Arm study of the endoluminal treatment of Abdominal Aortic Aneurysms using the Talent Endoluminal Spring Graft System
  Interventions: Device: Talent Endoluminal Spring Graft System

INTERVENTIONS:
Device: Talent Endoluminal Spring Graft System — Endovascular repair for patients with AAA who meet the inclusion criteria for the study

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the Talent Endoluminal Spring Graft System, an investigational device, to treat abdominal aortic aneurysms (AAA). The treatment population will include patients with an abdominal aortic aneurysm who meet the inclusion/exclusion criteria. All patients in the treatment population will undergo post-procedure follow-up evaluations at one (1), six (6), and 12 months and annually thereafter up to five (5) years post-procedure.

DETAILED DESCRIPTION:
Endovascular aneurysm repair (EVAR) offers certain advantages as compared to surgical repair of an abdominal aortic aneurysm. Known benefits associated with EVAR, as described in scientific literature, include minimally invasive procedure, shorter ICU and hospital stay, reduced blood loss, more rapid recovery, and reduced need for general anesthesia. Potential benefits that may be associated with use of the Talent device include reduced occurrence of endoleaks, therefore reduced subsequent re-interventions. The risks/complications known to occur to all patients undergoing AAA repair may include anesthetic complications, (e.g., aspiration), aneurysm enlargement, rupture, perforation or dissection, bleeding, arterial or venous thrombosis and/or pseudoaneurysm, arteriovenous fistula, hematoma or coagulopathy, bowel complications, cardiac complications, (e.g., arrhythmia, myocardial infarction, congestive heart failure, hypotension, hypertension), embolization (micro and macro) with transient or permanent ischemia or infarction, genitourinary complications, infection, neurologic complications, occlusion of device or native vessel, pulmonary/respiratory complications and renal complications.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who participate in this study must fulfill all of the following criteria.
* Subject is > 18 years of age.
* Subject is not pregnant, and, if female and of child-bearing potential, is practicing contraception.
* Subject has documented evidence of at least one patent internal iliac artery.
* Subject has an AAA that is dilated to > 4 cm in diameter.
* Subject has a proximal AAA neck (distance between the top of the aneurysm and the renal arteries) > 5 mm.
* Subject has a proximal aortic neck diameter > 14 mm and < 32 mm.
* Subject has an angle between the suprarenal aorta and the aneurysm <60o.
* Subject has renal arteries > 9 cm from the aortic bifurcation.
* Subject has proximal and distal iliac neck diameters > 8 mm and < 18 mm to accommodate stock devices. For those subjects whose proximal and distal iliac diameters are > 18 mm, custom devices with a variation in fixation diameters will be ordered from the manufacturer.
* Subject has a distal iliac neck length > 15 mm.
* Subject has signed informed consent.
* Subject will be available for follow-up for 12 months after the procedure.

Exclusion Criteria:

* Subjects who fulfill any of the following criteria may not participate in this study.
* Subject has patent internal iliac arteries that require graft extension to the external iliac arteries.
* Subject has one or more patent subrenal arteries with potential retrograde flow after stent-grafting.
* Subject has a dominant patent inferior mesenteric artery and an occluded or stenotic celiac and superior mesenteric artery.
* Subject has an aneurysm involving both internal iliac arteries.
* Subject has a lesion that cannot be crossed with a guide wire.
* Subject whose arterial access site cannot accommodate the delivery catheter.
* Subject has no distal vascular bed.
* Subject has systemic infection, or is suspected of having systemic infection.
* Subject has contraindications for use of contrast medium or anticoagulation drugs.
* Subject has received a previous stent in the subrenal aorta.
* Subject has an untreatable bleeding diathesis.
* Subject is in a hypercoagulable state.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2002-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodney A. White, M.D., Principal Investigator — Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Locations (1):
- LAC Harbor-UCLA Medical Center, Torrance, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: About 75 patients were screened for eligibility for enrollment in the study based on the inclusion/exclusion criteria. Participants were selected over a 7 year period between 2002 and 2008 and were made up of patients in the hospital, clinic patients as well as those referred from other clinics and facilities.
Groups:
- Talent Endoluminal Spring Graft System: All participants who were diagnosed with abdominal aortic aneurysms and who were eligible for enrollment as defined by the inclusion/exclusion criteria were screened. These patients included both high and low risk patients who signed a consent to participate in this Physician-sponsored IDE for the endoluminal treatment of their abdominal aneurysm using the Medtronic/Talent Stent Graft: Stent-graft for Abdominal Aortic Aneurysms.
Period: Overall Study
Arm/Group | Talent Endoluminal Spring Graft System
Started | 49 (75 patients were screened and a total of 49 were enrolled in the study.)
Completed | 18 (Eighteen (18) completed the study up to the 5 year followup.)
Not Completed | 31

BASELINE CHARACTERISTICS:
Groups:
- There Are no Study Arms.: All participants who were diagnosed with abdominal aortic aneurysms and who were eligible for enrollment as defined by the inclusion/exclusion criteria were screened. These patients included both high and low risk patients who signed a consent to participate in this Physician-sponsored IDE for the endoluminal treatment of their abdominal aneurysm using the Medtronic/Talent Stent Graft: Stent-graft for Abdominal Aortic Aneurysms.
Arm/Group | There Are no Study Arms.
Number analyzed (Participants) | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.64 (3.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 48
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 5
  White | 42
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 49

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Exclusion of Abdominal Aortic Aneurysm
Description: The safety and effectiveness of the endoluminal device was determined by the number participants with successful exclusion of the abdominal aortic aneurysm (AAA).
Time Frame: From the date of treatment assessed up to 5 years post treatment.
Measure: Number; unit: participants' AAA
Groups:
- Number of Successful Exclusion of Abdominal Aortic Aneurysms: The safety and effectiveness of the endoluminal device was determined by the number of abdominal aortic aneurysms (AAA) that were successfully excluded.
Arm/Group | Number of Successful Exclusion of Abdominal Aortic Aneurysms
Number analyzed (Participants) | 49
participants' AAA | 49

2. Secondary Outcome: Number of Participants With Successful Device Delivery and Deployment
Description: Delivery success is defined as the successful access of the vessel and insertion of the delivery sheath to the treatment site. Deployment success is defined as the advancement through the vasculature to the desired location and full deployment within 0.5 cm of the intended location. Aneurysm exclusion is achieved when there is no evidence of blood flow around or through the stent graft into the aneurysm or where there is an absence of contrast within the aneurysm sac.
Time Frame: From the date of treatment assessed up to 5 years post treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Number of Successful Device Delivery and Deployment: All participants who were diagnosed with abdominal aortic aneurysms and who were eligible for enrollment as defined by the entry criteria were screened. These patients included both high and low risk patients who signed a consent to participate in this Physician-sponsored IDE for the endoluminal treatment of their abdominal aneurysm using the Medtronic/Talent Stent Graft: Stent-graft for Abdominal Aortic Aneurysms.
Arm/Group | Number of Successful Device Delivery and Deployment
Number analyzed (Participants) | 49
Participants | 49

ADVERSE EVENTS:
Time Frame: From the data of treatment until the date of death from any event or the date of the adverse event assessed up to five years. Participants were followed for the duration of the study, an average of 5 years.
Groups:
- Talent Endoluminal Spring Stent Graft System: Endoluminal treatment of abdominal aortic aneurysms using the Medtronic/Talent Stent Graft: Stent-graft for all patients with abdominal aortic lesions who signed consent into this Physician - Sponsored IDE.
Arm/Group | Talent Endoluminal Spring Stent Graft System
All-Cause Mortality (participants affected / at risk) | 19/49
Serious Adverse Events (participants affected / at risk) | 29/49
Other Adverse Events (participants affected / at risk) | 4/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Talent Endoluminal Spring Stent Graft System (N=49)
Myocardial infarction (Cardiac disorders) | 2 (2)
Vessel Injury (Vascular disorders) | 1 (1)
Lung Cancer (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Congestive Heart Failure (Cardiac disorders) | 2 (2)
Endoleak (Vascular disorders) | 9 (9)
Ruptured AAA (Vascular disorders) | 1 (1) — 6 months post procedure
Ruptured TAA (Vascular disorders) | 1 (1) — 18 months post procedure
Renal Cancer (Renal and urinary disorders) | 1 (1)
Prostate cancer (Reproductive system and breast disorders) | 1 (1)
Stent Graft migration (Vascular disorders) | 2 (2) — At > 2 years post procedure
Stent Graft occlusion (Vascular disorders) | 3 (3) — At > 1 year post procedure
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Talent Endoluminal Spring Stent Graft System (N=49)
Hypertension (Vascular disorders) | 2 (2)
Peripheral Vascular Disease (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No